CLINICAL TRIAL: NCT02496403
Title: Buprenorphine and Substance Abuse Services for Prescription Opioid Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CN-13-1592-H; R01DA036603 (NIH)
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Opiate Substitution Treatment
Keywords: buprenorphine-naloxone combination; Suboxone; Buprenorphine; Substance Use; Behavioral intervention; Opioid partial agonist; medication assisted therapy; opioid addiction
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Medical Management (Experimental): Standard Medical Management (SMM) is a relatively brief (1.5 hour per week for 9 weeks), medically-focused behavioral intervention for opioid dependence. The experimental arm does not involve an investigational drug, device, or biologic.
  Interventions: Behavioral: Standard Medical Management (SMM)
- Intensive Outpatient Treatment (No Intervention): The Intensive Outpatient Treatment (IOT) arm is considered usual care and is a predominant model of care in specialty treatment. It incorporates psychosocial support, education, and relapse-prevention approaches and requires attendance at 12-step program. It is a group-based treatment, with individual counseling available as needed. During the initial, 3-week phase, treatment consists of 4-6 hours a day, 7 days a week. In weeks four through 9, treatment consists of 1.5 hours, four days each week. After 9 weeks, patients attend one-hour weekly group meetings for one year. Services include supportive therapy, psycho-education, relapse prevention, and family-oriented therapy. The program emphasis is on abstinence and is similar to many public and private intensive outpatient programs.

INTERVENTIONS:
Behavioral: Standard Medical Management (SMM) — SMM is designed to provide basic advice about opioid dependence and encouragement to adhere to treatment recommendations. Sessions provide support and monitoring of medication compliance, dose, withdrawal, adverse effects, and discussion of medical complications of opioid and other drug use. Early in treatment, the focus will be on helping patients adjust to the medications (e.g., monitoring withdrawal or other adverse symptoms, tolerating discomfort, curtailing illicit drug use, and referral to self-help). As treatment progresses, the practitioner may focus more on educating the patient about the social and behavioral factors perpetuating addiction and encourage behavioral and lifestyle change to support recovery.
  Arms: Standard Medical Management

SUMMARY:
This is a randomized trial of two group-based models of care for buprenorphine/naloxone (bup/nx) patients in Substance Use (SU) specialty treatment: Standard Medical Management (SMM) and Intensive Outpatient Treatment (IOT). The setting is a large outpatient SU treatment program, where a medical management model of care has not been empirically tested with bup/nx patients, and where a high prevalence of patients with co-occurring psychiatric and medical co-morbidities are treated. SSM includes brief weekly group-based visits consistent with previously studied medical models, and is drawn from primary care bup/nx research. IOT is a predominant model of care in specialty treatment, and incorporates psychosocial support, 12-step, educational and relapse-prevention based approaches. The investigators will recruit 300 adult patients inducted onto bup/nx, randomize them to either SMM or IOT, and conduct telephone follow-up interviews at 6 and 12 months. Study investigators will examine the impact of these treatment approaches on 90-day bup/nx adherence, opioid and SU abstinence, quality of life, and health care and societal costs. Further, investigators will examine whether the effect of IOT versus SMM on adherence and SU treatment outcomes is greater for those with medical or psychiatric co-morbidities. This innovative approach includes a focus on complex patients with psychiatric and medical co-morbidities in specialty care, adapting a care model previously only tested in primary care, a 12-month follow-up, no research-forced medication taper, an examination of health care and societal costs, and a combination of patient self-report and electronic medical record data. Through this approach, the proposed study will yield critically important findings on how best to treat complex prescription opioid dependent patients with an integrative behavioral services and medication treatment model in SU treatment.

DETAILED DESCRIPTION:
The study will contrast and compare the effectiveness and costs of two forms of behavioral SU treatment services for a total of 300 opioid dependent patients seeking bup/nx treatment at the Kaiser Sacramento Chemical Dependency Recovery Program (CDRP). The design is a between-groups clinical trial using blocked randomization to the two treatments (IOT and SMM) with analyses based on an intent-to-treat model.

Patients are recruited into the study and randomized after induction at the time of program intake. A full battery of background, concurrent status and diagnostic information will be collected at baseline, and repeated 6 and 12 months later to assess change in drug use, 30 day and 6-month abstinence, and quality of life at each point. The study will test for illicit drug use and presence of buprenorphine with random urinalysis throughout treatment. In addition to urinalysis, bup/nx adherence will be measured using prescription drug refills and self-report. Investigators will collect self-report of prescription opioid use and abstinence. Finally, the number and types of services received by during treatment will be available from the EMR.

Patients seeking bup/nx receive a 30-minute medical exam from a CDRP physician (e.g., for symptoms of alcohol or other drug withdrawal, hypertension, acute infections related to intravenous drug use, mental status, acute psychosis or suicidal tendencies) to assess appropriateness for bup/nx and discuss the treatment. After this initial evaluation, the induction is managed by the clinic nurse, in consultation with a clinic physician. Induction follows the standard of care, and occurs over 2-3 days. The average daily dose of bup/nx ranges from 12-24mg, but is typically 16 mg.

After induction, the patient will be scheduled for an intake interview for admission into the treatment program. Following the intake session, a research staff member will describe the study and assess eligibility criteria. For patients who agree to participate, the research associate will proceed to enroll the patient in a private room. During enrollment/baseline appointment, the research associate will obtain informed consent and administer a baseline questionnaire using a laptop computer (see below). Patients will then be randomized to either the IOT or SMM arm using a block randomization procedure which will ensure that equal numbers of patients will be assigned to each treatment arm. Patients unwilling or unable to be randomized will meet with the intake therapist and treated in the standard manner designated by the treatment program's regular intake counselors, and will not be part of the study.

At baseline, following recruitment and consent, participants will complete a computerized interview in a private place at the CDRP (with a research associate available for any computer or content questions). A full battery of background, physical and mental health and SU disorder information will be collected.

Study investigators will conduct two follow-up telephone interviews whether or not patients complete the CDRP treatment program. At the follow-up, participants will be reminded of the study and permission to conduct the interview will be obtained verbally. Interviews will be conducted at 6 and 12 months by research staff with the same baseline measures to assess treatment adherence, substance use and abstinence, and quality of life. Also, patients will be asked to present at the CDRP within 48 hours of the 6 and 12 month interviews for a urine test and additional brief questions on drug use.

ELIGIBILITY:
Inclusion Criteria:

* inducted for buprenorphine/naloxone treatment at the Sacramento CDRP
* diagnosis of opioid dependence
* English speaking
* Willing and able to be randomized to treatment arm

Exclusionary criteria:

* dementia
* mental retardation
* actively psychotic or suicidal
* medically unstable
* using opioids
* pregnant women
* inducted on bup/nx for chronic pain
* inducted on bup/nx for detoxification purposes only
* enrolled in DDIOP, residential treatment or day treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Adherence to buprenorphine/naloxone using MPR | 90-day
  Buprenorphine/naloxone adherence will be measured using KPNC's pharmacy database. Adherence will be based on prescription refills and calculated using Medication Possession Ratio methods, similar to other published KPNC studies which have measured adherence as a key outcome variable. Adherence will be defined as the patient having medication available on 80% or more of the 90 day period-that is, an MPR of .8 or higher.
Abstinence using ASI | 6 months
  We use composite measures from the Addiction Severity (ASI) index to examine 30 day abstinence outcomes for opioids and other substances (marijuana, cocaine, methamphetamine and other stimulants, hallucinogens, barbiturates, tranquilizers, inhalants, hallucinogens).
Health care utilization costs using ICER | 12 months
  Substance use treatment utilization data (number of visits, number of days in treatment), as well as general health care utilization data (inpatient, outpatient, and ER) will be collected using the electronic medical record. In addition, health care utilization outside Kaiser will be assessed and used to create composite measure of health care utilization costs. The incremental cost-effectiveness ratio (ICER) will be calculated for each additional unit of outcome as the ratio of difference in costs between the two arms divided by the difference in outcome.
Adherence to buprenorphine/naloxone using drug testing | 90-day
  Urine tests will be performed weekly during treatment. If 80% of test results within the 90-day period are positive during the 90 day period, we will consider the patient to be adherent to treatment.
Abstinence using ASI | 12 months
  We use composite measures from the Addiction Severity (ASI) index to examine 30 day abstinence outcomes for opioids and other substances (marijuana, cocaine, methamphetamine and other stimulants, hallucinogens, barbiturates, tranquilizers, inhalants, hallucinogens).

SECONDARY OUTCOMES:
Chronic Pain using the pain Interference scale | 6 months
  The severity of chronic pain and the degree to which it interferes with every day life will be measured using the PROMIS Pain Interference scale.
Quality of Life using PROMIS Global Health scale | 6 months
  Quality of life will be assessed by the PROMIS Global Health scale, which measures satisfaction with physical health, psychological health, and social relationships.
Mental health using PHQ-9 | 6 months
  Psychiatric problem severity will be measured by the PHQ-9, a 9-item measure of depression and anxiety symptoms.
Chronic Pain using the pain Interference scale | 12 months
  The severity of chronic pain and the degree to which it interferes with every day life will be measured using the PROMIS Pain Interference scale.
Mental health using PHQ-9 | 12 months
  Psychiatric problem severity will be measured by the PHQ-9, a 9-item measure of depression and anxiety symptoms.
Quality of Life using PROMIS Global Health scale | 12 months
  Quality of life will be assessed by the PROMIS Global Health scale, which measures satisfaction with physical health, psychological health, and social relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Campbell, PhD, Principal Investigator — Kaiser Permanente Division of Research
Locations (1):
- Kaiser Sacramento Chemical Dependency Recovery Program, Sacramento, California, United States

REFERENCES:
- [Background] Miller C, Dadoo R, Kooser RG, Gorse J. Electron spin resonance studies under dynamic mobile phase conditions on chemically modified silica. J Chromatogr. 1988 Dec 23;458:255-66. doi: 10.1016/s0021-9673(00)90569-7. PMID 2853172
- [Background] International Symposium on Electroanalysis in Biochemical, Environmental and Industrial Sciences. Loughborough, UK, 11-14 April, 1989. Proceedings. Analyst. 1989 Dec;114(12):1517-705. doi: 10.1039/an9891401517. No abstract available. PMID 2633651
- [Background] Haddad MS, Zelenev A, Altice FL. Integrating buprenorphine maintenance therapy into federally qualified health centers: real-world substance abuse treatment outcomes. Drug Alcohol Depend. 2013 Jul 1;131(1-2):127-35. doi: 10.1016/j.drugalcdep.2012.12.008. Epub 2013 Jan 17. PMID 23332439
- [Background] Stein BD, Gordon AJ, Sorbero M, Dick AW, Schuster J, Farmer C. The impact of buprenorphine on treatment of opioid dependence in a Medicaid population: recent service utilization trends in the use of buprenorphine and methadone. Drug Alcohol Depend. 2012 Jun 1;123(1-3):72-8. doi: 10.1016/j.drugalcdep.2011.10.016. Epub 2011 Nov 16. PMID 22093488
- [Background] Soeffing JM, Martin LD, Fingerhood MI, Jasinski DR, Rastegar DA. Buprenorphine maintenance treatment in a primary care setting: outcomes at 1 year. J Subst Abuse Treat. 2009 Dec;37(4):426-30. doi: 10.1016/j.jsat.2009.05.003. Epub 2009 Jun 23. PMID 19553061
- [Background] Manchikanti L, Fellows B, Ailinani H, Pampati V. Therapeutic use, abuse, and nonmedical use of opioids: a ten-year perspective. Pain Physician. 2010 Sep-Oct;13(5):401-35. PMID 20859312
- [Background] Kenan K, Mack K, Paulozzi L. Trends in prescriptions for oxycodone and other commonly used opioids in the United States, 2000-2010. Open Med. 2012 Apr 10;6(2):e41-7. Print 2012. PMID 23696768
- [Background] Graybill JR. Histoplasmosis and AIDS. J Infect Dis. 1988 Sep;158(3):623-6. doi: 10.1093/infdis/158.3.623. No abstract available. PMID 3045214
- [Background] Presl J. [Bioactive and immunoreactive gonadotropins]. Cesk Gynekol. 1986 Jun;51(5):354-8. No abstract available. Czech. PMID 3087632
- [Background] Sitges-Serra A, Alonso M, de Lecea C, Gores PF, Sutherland DE. Pancreatitis and hyperparathyroidism. Br J Surg. 1988 Feb;75(2):158-60. doi: 10.1002/bjs.1800750224. PMID 3280087
- [Background] Heinen E, Braun M, Louis E, Cormann N, Tsunoda R, Kinet-Denoel C, Lesage F, Simar LJ. Interactions between follicular dendritic cells and lymphoid cells. Adv Exp Med Biol. 1988;237:181-4. doi: 10.1007/978-1-4684-5535-9_26. No abstract available. PMID 2978198
- [Background] Kitagawa T, Pitot HC. Immunohistochemical demonstration of serine dehydratase in rat liver. Am J Pathol. 1975 Feb;78(2):309-18. PMID 163593
- [Background] Kuehn BM. Opioid prescriptions soar: increase in legitimate use as well as abuse. JAMA. 2007 Jan 17;297(3):249-51. doi: 10.1001/jama.297.3.249. No abstract available. PMID 17227967
- [Background] Coben JH, Davis SM, Furbee PM, Sikora RD, Tillotson RD, Bossarte RM. Hospitalizations for poisoning by prescription opioids, sedatives, and tranquilizers. Am J Prev Med. 2010 May;38(5):517-24. doi: 10.1016/j.amepre.2010.01.022. PMID 20409500
- [Result] Oakey RE. Steroid sulphatase deficiency. J Endocrinol. 1987 Mar;112(3):341-3. doi: 10.1677/joe.0.1120341. No abstract available. PMID 3470422
- See also: Centers for Disease Control and Prevention. Vital signs: Overdoses of prescription opioid pain relievers --- United States, 1999--2008. MMWR. 2011;60(43):1487-1492. — http://www.cdc.gov/mmwr/preview/mmwrhtml/mm6043a4.htm?s_cid=mm6043a4_w.